CLINICAL TRIAL: NCT05388500
Title: Protocol for Herceptin as Adjuvant Therapy With Reduced Exposure to Chemotherapy, a Randomised Comparison of Trastuzumab vs Trastuzumab+Paclitaxel in Women With HER2-positive Early Breast Cancer Receiving Neoadjuvant Treatment
Brief Title: Protocol for Herceptin as Adjuvant Therapy With Reduced Exposure to Chemotherapy (PHARE-C)
Acronym: PHARE-C
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-008
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Paclitaxel + Trastuzumab) (Active Comparator)
  Interventions: Drug: Paclitaxel + Trastuzumab
- Group B (Trastuzumab) (Experimental)
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Paclitaxel + Trastuzumab — Regarding neoadjuvant treatment :
  - 9 to 12 weeks of neoadjuvant treatment Trastuzumab IV (8mg/kg loading dose followed by 6 mg/kg maintenance dose) or SubCutaneous (SC) (600mg fixed dose) every 3 weeks + weekly Paclitaxel IV : 80 to 90 mg/m2
  Regarding adjuvant treatment patients will receive one of the following anti-HER2 therapy following the current standard to complete 1 year of anti-HER2 therapy in total :
  * in case of pCR : patient will receive trastuzumab
  * in case of non pCR : patients will receive trastuzumab emtansine (T-DM1)
  Arms: Group A (Paclitaxel + Trastuzumab)
Drug: Trastuzumab — Regarding neoadjuvant treatment :
  - 9 to 12 weeks of neoadjuvant treatment Trastuzumab IV (8mg/kg loading dose followed by 6 mg/kg maintenance dose) or SC (600mg fixed dose) every 3 weeks
  Regarding adjuvant treatment patients will receive one of the following anti-HER2 therapy following the current standard to complete 1 year of anti-HER2 therapy in total :
  * in case of pCR : patient will receive trastuzumab
  * in case of non pCR : patients will receive trastuzumab emtansine (T-DM1)
  Arms: Group B (Trastuzumab)

SUMMARY:
RATIONALE: According to previous results from PHARE study, a subgroup of patients with low-risk cancer (< 3 cm) without axillary lymph node involvement or small (< 2 cm) with minimal lymph node involvement (1 positive node) presented low risk of recurrence. Maintaining chemotherapy in this subgroup could cause toxicity and it is not yet known whether giving trastuzumab as monotherapy in neoadjuvant setting is as effective as giving trastuzumab combined with paclitaxel in patients with low risk early breast cancer.

PURPOSE: This randomized phase III trial is studying trastuzumab as monotherapy in neoadjuvant setting to see if this treatment regimen is as efficient compared to trastuzumab combination with paclitaxel chemotherapy in treating women with low risk (tumor size< 3 cm, N0) early breast cancer.

DETAILED DESCRIPTION:
PHARE-C is an open-label, randomized, phase III, non-inferiority trial, that will recruit patients with human epidermal growth factor receptor 2 (HER2)-positive early breast cancer to allow for comparison of neoadjuvant treatment with paclitaxel plus trastuzumab versus trastuzumab as monotherapy.

Non-inferiority between the two treatment arms will be evaluated in terms of time to progression as primary objective. Treatment tolerance and cardiac toxicity will be assessed as secondary objectives.

In case of non pCR, a rescue by Trastuzumab emtansine (T-DM1) is planned to control the survival outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast, nonmetastatic disease and non operated tumor
* Without suspicious axillary nodes
* Tumor size < 30 mm
* Eligibility to receive a weekly paclitaxel based chemotherapy for this cancer
* Left Ventricular Ejection Fraction (LVEF) obtained and > 50% as measured by echocardiography (Simpson method) or multigated acquisition scan (MUGA) at 3 months (-/+ 1 month)
* Overexpression of HER-2 in the invasive component of the primary tumor as indicated by one of the following:

  3+ by immunohistochemistry (IHC) 2+ by IHC and confirmation by fluorescent in situ hybridization (FISH) or chromogenic in situ hybridization (CISH)
* With signed Informed consent

Exclusion Criteria:

* Previous anti-HER2 treatment (except for HERCEPTIN)
* Cardiac disease or other medical conditions preventing trastuzumab administration
* Known allergy to trastuzumab, murine proteins or other excipients
* Pregnant or breastfeeding women
* Patients that are not able to comply to the protocol assessments for geographic, social or psychological reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 800 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2030-12-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
Time to progression | up to 5 years
  Time from the date of randomization to the date of progression

SECONDARY OUTCOMES:
Cardiac toxicity | up to 5 years
  defined by Ventricular Ejection Fraction measure according to the technique used, clinical examination or any other appropriate exams
Treatment toxicity | up to 5 years
  Adverse Event and Serious Adverse Event due to trastuzumab or paclitaxel graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Total pathological Complete Response (tpCR) | through surgery completion, an average of 12 weeks
  Defined by complete absence of cancerous cells in breast, axillary lymph node chain and/or axillary sentinel lymph node (ypT0/is) in excised tissues
Breast pathological Complete Response (bpCR) | through surgery completion, an average of 12 weeks
  Defined by complete absence of cancerous cells in breast (ypT0/is, ypN0) in excised tissues
Distant metastasis Free Survival | up to 5 years
  Time from the date of randomization to the date of 1st metastasis
Overall Survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Xavier PIVOT, MD, PhD, Study Chair — Institut de cancérologie Strasbourg Europe